CLINICAL TRIAL: NCT06195215
Title: The Effect of Peer Counseling Initiative Applied to First Year Nursing Students in the Orientation Process on Their Perception of Nursing Image
Brief Title: The Effect of Peer Counseling on Nursing Image
Acronym: peer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, SÜMEYYE KAYA KOCAGİL, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: SKaya_002
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Nursing
Keywords: nursing image; nursing student; orientation; peer education
MeSH Terms: conditions — Orientation, Spatial

STUDY DESIGN:
Intervention Model Description: The research will be conducted in a single-centre, parallel group, randomised controlled pretest-posttest design.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peer counselling (Experimental): * Does not have any cognitive, affective and verbal problems that prevent communication
  * It is planned to include nursing students with an Image Scale for Nursing Profession score of 143 and lower.
  * The peer counselling process related to nursing image was applied to this group by 1 senior nursing student for 1 hour a week for 7 weeks. Before and immediately after the 7-week period, the nursing image scale is applied.
  Interventions: Other: Peer Counselling
- Control (No Intervention): * Does not have any cognitive, affective and verbal problems that prevent communication
  * It is planned to include nursing students with an Image Scale for Nursing Profession score of 143 and lower.
  * No peer counselling process is applied to this group. Seven weeks after the first data collection, the final data are collected for the second time using the nursing image scale.

INTERVENTIONS:
Other: Peer Counselling — 7 weeks peer counselling process will be carried out.
  Arms: peer counselling

SUMMARY:
The aim of this randomised controlled study was to examine the effect of peer counselling on first-year nursing students' perceptions of nursing image in orientation processes.The H0 hypothesis of the study is that there is no statistical difference between the scores of the image scale towards nursing between the experimental and control groups after the peer-assisted orientation process.

DETAILED DESCRIPTION:
In the study, pre-test data will be collected from the first year students enrolled in the school by using the 'Sociodemographic Data Form' and the 'Image Scale for Nursing Profession'. According to the pre-test results, 108 first-year nursing students who scored 143 points or less from the Image Scale for Nursing Profession will be determined by an independent statistical expert. These students will then be assigned to the experimental (n=54) and control (n=54) groups by simple randomisation method. The students in the intervention group will be randomly grouped with 27 senior nursing students who voluntarily agree to participate in the project to provide peer counseling, and one senior student will counsel 2 first-year students. A 7-week counseling process of 1 hour per week will be applied to 54 students in the intervention group. The research will be finalised by applying the post-test to the control and intervention groups immediately after the intervention.

ELIGIBILITY:
Inclusion Criteria:

The experimental and control group to be included in the study

* Continuing their education in the first year of Mersin University Faculty of Nursing in the 2023-2024 Academic Year,
* Willing to participate in the study voluntarily, signing the informed consent form/written consent form,
* Does not have any cognitive, affective and verbal problems that prevent communication
* It is planned to include nursing students with an Image Scale for Nursing Profession score of 143 and lower.

Exclusion Criteria:

The experimental and control group to be excluded in the study

* Do not wish to participate as a volunteer, do not sign the informed consent form/written consent form
* Have a problem that prevents them from communicating cognitively, emotionally and verbally,
* It is planned to exclude nursing students with an Image Scale for Nursing Profession score of 143 and higher from the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Nursing image scores evaluated using Image Scale for Nursing Profession | Before the intervention, Immediately after the intervention.
  Scores ranging from 42 to 210. It is a 5-point Likert type scale and consists of 42 items. It is evaluated between 5 'strongly agree' and 1 'strongly disagree'. Items 8, 14, 15, 17, 18, 20, 21, 21, 22, 23, 23, 24, 25, 26, 28, 29 and 31 are reverse coded. As the score obtained from the scale increases, nurses' perception of professional image increases positively. Scale 143-109 points indicate medium level image, 108 and below indicate low level nursing image.

CONTACTS AND LOCATIONS:
Overall Officials: Sümeyye Kaya Kocagil, Master, Principal Investigator — Mersin Üniversity
Locations (1):
- Turkey, Mersin Üniversity, Mersin, Turkey (Türkiye)

REFERENCES:
- [Background] Apaydin Cirik V, Gul U, Aksoy B. The image of nursing among nursing and other healthcare professional university students: A mixed-method study. Nurse Educ Pract. 2022 Feb;59:103293. doi: 10.1016/j.nepr.2022.103293. Epub 2022 Jan 12. PMID 35066255